CLINICAL TRIAL: NCT04574921
Title: ALZLIGHT Pilot: Study on Safety, Feasibility and Neural Activation of Non-Invasive Light Therapy System
Brief Title: Study on Safety, Feasibility and Neural Activation of Non-Invasive Light Therapy System
Acronym: ALZLIGHT Pilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zealand University Hospital (Other)
Collaborators: Technical University of Denmark (Other); University of Copenhagen (Other); OptoCeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: REG-085-2020
Record Dates: First submitted 2020-08-27; First posted 2020-10-05 (Actual); Last update posted 2022-12-13 (Actual); Status verified 2022-12

CONDITIONS: Alzheimer Disease
Keywords: Gamma entrainment; 40 Hz; Invisible Spectral Flicker; LED; Light Therapy; Brain stimulation; Gamma oscillations; Gamma induction
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active (Experimental): Exposure to LTS device set to 40 Hz invisible spectral flicker for 1 hour a day for consecutive days
  Interventions: Other: Light Therapy System (LTS): Active setting
- Sham (Sham Comparator): Exposure to LTS device set to continues color matched white light for 1 hour a day for consecutive days
  Interventions: Other: Light Therapy System (LTS): Sham setting

INTERVENTIONS:
Other: Light Therapy System (LTS): Active setting — Exposure for 1 hour á day for consecutive days.
  Arms: Active
Other: Light Therapy System (LTS): Sham setting — Exposure for 1 hour á day for consecutive days.
  Arms: Sham

SUMMARY:
Induction of neural oscillations by flickering light is a well established method used for diagnostic of various neural diseases.

Recent studies in mice have shown promising results indicating that induction of gamma oscillation at 40 Hz leads to a reduction in amyloid-β and tau in mice models of Alzheimer's disease. This study will use flickering light to induce 40 Hz gamma oscillation as the previously mentioned studies.

In the study subject will be exposed to invisible spectral flickering light (active setting) or continuous non-flickering white light (sham setting) for 1 hour each day. The sham setting is a high quality sham intervention as subjects will be blinded to the setting, both appears as white light.

As this is the first trial, the focus will be on 1) safety of the intervention 2) feasibility of the proposed intervention time and method 3) indication of efficacy.

In stage 1 of the trial 4 age-matched subjects with no Alzheimer's disease will be recruited and be exposed for 1 week. In stage 2 10 patients with Alzheimer's disease will be recruited and exposed for 6 consecutive weeks.

DETAILED DESCRIPTION:
Induction of neural oscillations by flickering light is a well established method used for diagnostic of various neural diseases (5,6).

Recent studies in mice have shown promising results indicating that induction of gamma oscillation at 40 Hz leads to a reduction in amyloid-β an tau in mice models of Alzheimer's disease (1-4). This study will use flickering light to induce 40 Hz gamma oscillation as the previously mentioned studies.

This study will utilize a novel way of masking the light by alternating the spectral composition of a white light, rendering the flicker invisible to the conscience perception while still entraining 40 Hz oscillations in the brain.

In the study subject will be exposed to invisible spectral flickering light (active setting) or continuous non-flickering white light (sham setting) for 1 hour each day. The sham setting is a high quality sham intervention as subjects will be blinded to the setting, both appears as white light.

As this is the first trial, the focus will be on 1) safety of the intervention 2) feasibility of the proposed intervention time and method 3) indication of efficacy.

In stage 1 of the trial 4 age-matched subjects with no Alzheimer's disease will be recruited and be exposed for 1 week. In stage 2 10 patients with Alzheimer's disease will be recruited and exposed for 6 consecutive weeks. Following the 6 weeks of intervention the subject will have 6 weeks of no intevention and assesed agian.

ELIGIBILITY:
Inclusion Criteria:

* Adult competent persons able to understand the nature of the study and give written informed consent.
* Stage I: Healthy elderly subject.
* Stage II: Diagnosed with probable mild to moderate AD based on NIA-AA diagnostic criteria.
* Age >55 years and <80 years. Females must be post-menopausal.
* Fluent in Danish
* > 8 year of normal school education
* Pass a colour-blindness test (Ishihara colour test)
* Have visual and auditory capabilities, and language skills necessary for neuropsychological testing.
* Furthermore, subjects must have a person, hereafter named designated caregiver, who is available to the participant and can provide the necessary assistance with using the LTS device and Actigraph wearable at home and can assist with clinic visits and other practical issues.

Exclusion Criteria:

* Profound visual impairment provided correction with spectacles, if needed.
* Significant abnormalities related to important parts of the brain e.g. the visual system, pre-frontal cortex or hippocampus, or relevant lesions detected by MRI.
* Prior history of significant diseases related to the visual system or the brain.
* Medication Any patient using antiepileptic drugs, neuromodulating drugs or high dose of sedatives will be excluded.
* Prior history of substance abuse within the past 2 years.
* Any significant systemic illness or unstable medical condition, which could lead to difficulty complying with the protocol.

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-07-12 (Actual); Study Completion 2022-07-12 (Actual)

PRIMARY OUTCOMES:
Stage I: Feasibility / Compliance assesment | After 1 week of intervention
  • The compliance of the LTS intervention will be measured by the amount of time (in minutes) of device use per day.
Stage I: Usability Assessment: | After 1 week of intervention
  • Usability report on use of device during intervention in the subject's home based on device speciffic questionnaire / structured interviews
Stage I: Safety Assessment. Evaluation of Adverse Events related to the LTS intervention. | After 1 week of intervention
  • Safety assessment will be done by collection of all types of adverse events and categorization into severity and relationship to LTS treatment.
Stage II: Feasibility / Compliance assesment | After 6 weeks of intervention and subsequent 6 weeks of no intervention
  • The compliance of the LTS intervention will be measured by the amount of time (in minutes) of device use per day.
Stage II: Safety Assessment. Evaluation of Adverse Events related to the LTS intervention. | After 6 weeks of intervention and subsequent 6 weeks of no intervention
  • Device- and procedure-related adverse events (DR/PR-AEs) including serious AEs (SAEs) occurring at any time during the trial

SECONDARY OUTCOMES:
Stage II: Induction of gamma ocsillations | Changes from baseline to 6 and 12 weeks
  • The effect of the LTS intervention will be measured by the amount of 40 Hz SSVEP response during treatment
Stage II: Connectivity meassures in resting-state functional MRI | Changes from baseline to 6 and 12 weeks
  • rs-fMRI Connectivity: Change from baseline in correlations between cortical regions at 6 weeks
Stage II: Connectivity meassures in EEG | Changes from baseline to 6 and 12 weeks
  • EEG Connectivity: Change from baseline in correlations between cortical regions at 6 weeks

OTHER OUTCOMES:
Stage II: Changes in cognition: | Changes from baseline to 6 and 12 weeks
  • Changes in cognition meassured by the ADAS Cog Plus EF & FA neuropsychological test. Score from 0 to 200
Stage II: Changes in cognition: | Changes from baseline to 6 and 12 weeks
  • Changes in cognition meassured by the Trailmaking A&B score from 0 to 1200 seconds
Stage II: Changes MR spectroscopy | Changes from baseline to 6 and 12 weeks
  • Chance from baseline in brain metabolism at 6 weeks
Stage II: Changes MR Perfusion | Changes from baseline to 6 and 12 weeks
  • Chance from baseline in perfusion meassured by Arterial Spin Labelling at 6 weeks
Stage II: Changes MR volumemetry | Changes from baseline to 6 and 12 weeks
  • Chance from baseline in structural volume of neural structures at 6 weeks
Stage II: Changes in Sleep Quality: | Changes from baseline to 6 and 12 weeks
  • Actigraphy: To assess changes in sleep patterns
Stage II: EEG spectral features: | Changes from baseline to 6 and 12 weeks
  • rs-EEG fourier power: To assess changes in spectral features

CONTACTS AND LOCATIONS:
Locations (1):
- Zealand University DK34197393, Roskilde, Region Sjælland, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Adaikkan C, Middleton SJ, Marco A, Pao PC, Mathys H, Kim DN, Gao F, Young JZ, Suk HJ, Boyden ES, McHugh TJ, Tsai LH. Gamma Entrainment Binds Higher-Order Brain Regions and Offers Neuroprotection. Neuron. 2019 Jun 5;102(5):929-943.e8. doi: 10.1016/j.neuron.2019.04.011. Epub 2019 May 7. PMID 31076275
- [Background] Adaikkan C, Tsai LH. Gamma Entrainment: Impact on Neurocircuits, Glia, and Therapeutic Opportunities. Trends Neurosci. 2020 Jan;43(1):24-41. doi: 10.1016/j.tins.2019.11.001. Epub 2019 Dec 10. PMID 31836315
- [Background] Iaccarino HF, Singer AC, Martorell AJ, Rudenko A, Gao F, Gillingham TZ, Mathys H, Seo J, Kritskiy O, Abdurrob F, Adaikkan C, Canter RG, Rueda R, Brown EN, Boyden ES, Tsai LH. Gamma frequency entrainment attenuates amyloid load and modifies microglia. Nature. 2016 Dec 7;540(7632):230-235. doi: 10.1038/nature20587. PMID 27929004
- [Background] Martorell AJ, Paulson AL, Suk HJ, Abdurrob F, Drummond GT, Guan W, Young JZ, Kim DN, Kritskiy O, Barker SJ, Mangena V, Prince SM, Brown EN, Chung K, Boyden ES, Singer AC, Tsai LH. Multi-sensory Gamma Stimulation Ameliorates Alzheimer's-Associated Pathology and Improves Cognition. Cell. 2019 Apr 4;177(2):256-271.e22. doi: 10.1016/j.cell.2019.02.014. Epub 2019 Mar 14. PMID 30879788
- [Background] Herrmann CS. Human EEG responses to 1-100 Hz flicker: resonance phenomena in visual cortex and their potential correlation to cognitive phenomena. Exp Brain Res. 2001 Apr;137(3-4):346-53. doi: 10.1007/s002210100682. PMID 11355381
- [Background] Kasteleijn-Nolst Trenite D, Rubboli G, Hirsch E, Martins da Silva A, Seri S, Wilkins A, Parra J, Covanis A, Elia M, Capovilla G, Stephani U, Harding G. Methodology of photic stimulation revisited: updated European algorithm for visual stimulation in the EEG laboratory. Epilepsia. 2012 Jan;53(1):16-24. doi: 10.1111/j.1528-1167.2011.03319.x. Epub 2011 Nov 16. PMID 22091642
- See also: Carstensen M et al. 40 Hz invisible spectral flicker and its potential use in Alzheimer's light therapy treatment. Proc. SPIE 11221, Mechanisms of Photobiomodulation Therapy XV, 112210L (11 March 2020) — https://doi.org/10.1117/12.2544338